CLINICAL TRIAL: NCT06663943
Title: A Prospective, Single-Center, Open-Label, Randomized Clinical Study on the Treatment of Pemphigus With a Novel Humanized CD38 Monoclonal Antibody (CM313)
Brief Title: A Randomized Study on Pemphigus Treatment With Humanized CD38 Antibody CM313.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chao Ji (Other)
Responsible Party: Sponsor-Investigator, Chao Ji, Chief Physician, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FirstAHFujian456
Record Dates: First submitted 2024-10-14; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Pemphigus Disease; Pemphigus Vulgaris (PV)
Keywords: Pemphigus; CD38; CM313; Autoantibodies
MeSH Terms: conditions — Pemphigus | interventions — Glucocorticoids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM313 (SC)、Glucocorticoid (Prednisone) (Experimental): Patients in the experimental group receive CM313 in combination with steroid therapy, with CM313 600mg (4ml/vial) administered subcutaneously at 0 and 1/2 weeks, followed by administration every 6 months or as determined by clinical assessment; subcutaneous injections are performed by doctors from this hospital, and patients are treated according to the normal outpatient diagnostic and treatment process; participants can have DSG antibody testing for free, and doctors will regularly follow up with patients by phone to monitor changes in their condition; the observation and follow-up period is 56 weeks.
  Interventions: Drug: CM313 (SC)
- Glucocorticoid (prednisone), azathioprine (Active Comparator): Patients in the control group receive azathioprine in combination with steroid therapy. The dosage of azathioprine (AZA) is adjusted based on the activity of thiopurine methyltransferase (TPMT), and TPMT activity should be measured before the administration of azathioprine. For individuals with normal TPMT activity, it is recommended to use AZA at a dosage of 2.0-3.0 mg·kg/d; for patients with TPMT enzyme mutations, it is recommended to use AZA at a dosage of 0.5-1.5 mg·kg/d. The initial treatment dose is suggested to be 50 mg AZA per day; the dose can be increased to the optimal dosage based on TPMT activity.
  Interventions: Drug: Glucocorticoids

INTERVENTIONS:
Drug: CM313 (SC) — CM313 is an anti-CD38 monoclonal antibody that can help pemphigus patients systematically treat rapid glucocorticoid reduction. It has been proven to have good safety in non-clinical studies and is suitable for human studies
  Arms: CM313 (SC)、Glucocorticoid (Prednisone)
Drug: Glucocorticoids — Patients in the control group receive azathioprine in combination with steroid therapy.
  Arms: Glucocorticoid (prednisone), azathioprine

SUMMARY:
Pemphigus is characterized by the presence of IgG antibodies that lead to the loss of keratinocyte adhesion, resulting in blister formation. The etiology of pemphigus antibodies is multifactorial, involving immune dysregulation, genetic predisposition, and potential viral triggers. CD38, a multifunctional transmembrane glycoprotein, plays a crucial role in B-cell maturation and function. CM313, a novel humanized monoclonal antibody targeting CD38, has shown promise in clinical trials for autoimmune diseases, including refractory/relapsed multiple myeloma (RRMM), systemic lupus erythematosus (SLE), and immune thrombocytopenia (ITP). By binding to CD38 on B cells, CM313 modulates B-cell activation, proliferation, and differentiation, potentially reducing the production of autoantibodies, such as those against desmogleins 1/3 in pemphigus. Preclinical studies have demonstrated that CM313 effectively inhibits CD38 enzymatic activity through antibody-dependent cellular cytotoxicity (ADCC), complement-dependent cytotoxicity (CDC), antibody-dependent cellular phagocytosis (ADCP), and Fc-mediated apoptosis. The long-term modulation of B-cell-mediated immune responses by CM313, through the depletion of both short-lived and long-lived plasma cells, suggests a novel therapeutic strategy for pemphigus by targeting the production of pathogenic autoantibodies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnostic criteria for pemphigus, including:

   ①Clinical manifestations: The presence of flaccid bullae and vesicles on the skin that are prone to rupture.

   Formation of persistent erosions following the rupture of bullae and vesicles. Vesicles or erosions on mucous membranes.

   ②Positive Nikolsky's sign.

   Histopathological findings:

   Intercellular acantholysis within the epidermis or epithelium, leading to the formation of bullae and vesicles.

   ③Immunodiagnostic indicators: Direct immunofluorescence (DIF) showing IgG and/or complement deposition between epidermal (or epithelial) cells in lesional or perilesional normal skin； Indirect immunofluorescence (IIF) detecting anti-epithelial cell antibodies in serum；Enzyme-linked immunosorbent assay (ELISA) detecting anti-desmoglein antibodies in serum.

   Diagnosis is confirmed with at least one clinical manifestation plus one of the histopathological or immunodiagnostic indicators, or at least two clinical manifestations plus two immunodiagnostic indicators.
2. Adult patients aged between 18 and 80 years.
3. Patients with moderate to severe generalized or vegetans pemphigus, as determined by a Pemphigus Disease Area Index (PDAI) score of 9-24 for moderate and ≥25 for severe.
4. Patients receiving CM313 treatment for the first time, including those with inadequate response to prior rituximab or other treatments.
5. Patients who have provided informed consent, agree to the treatment plan, and are willing to participate in follow-up assessments.

Exclusion Criteria:

1. Patients diagnosed with proliferative pemphigus, paraneoplastic pemphigus, or other autoimmune bullous diseases.
2. Patients who have received intravenous cyclophosphamide, plasmapheresis, or immunoadsorption treatment within 8 weeks prior to randomization.
3. Patients who have undergone rituximab or other B-cell targeted therapies within 3 months prior to randomization.
4. Patients with known active HIV, hepatitis B, or hepatitis C infection, as indicated by positive serology.
5. Patients with any known active infection (excluding fungal infections of the skin and nail beds).
6. Pregnant or breastfeeding women, and women of childbearing potential who are planning to become pregnant.
7. Other exclusions include:

   * Patients with known hypersensitivity to anti-CD38 monoclonal antibodies or excipients, or those who have previously received anti-CD38 monoclonal antibody therapy with inadequate response.
   * Patients with a history of thrombotic or embolic events or extensive severe bleeding within 6 months prior to the first dose of the study drug, such as hemoptysis, severe upper gastrointestinal bleeding, intracranial hemorrhage, sepsis, or irregular bleeding.
   * Patients who have participated in any other investigational drug study (including vaccine studies) or have been exposed to other investigational drugs within 4 weeks or 5 half-lives (whichever is longer) before the first dose of the study drug.
   * Patients who have received live vaccines within 4 weeks prior to the first dose of the study drug or who plan to receive any live vaccines during the study.
   * Patients who have undergone allogeneic stem cell transplantation or organ transplantation.
   * Patients with a significant medical history within the past 6 months that, in the opinion of the investigator, poses a risk to the patient's safety during the study or may affect the analysis of safety or efficacy. This includes major clinical histories such as cardiovascular events (e.g., acute myocardial infarction, heart failure, unstable angina, serious arrhythmias, etc.), New York Heart Association (NYHA) Class III-IV heart failure, poorly controlled diabetes, peptic ulcers, liver or kidney dysfunction, and various connective tissue diseases.
   * Patients with a history of malignant tumors within the past 5 years (excluding completely cured in situ cervical cancer and non-melanoma skin squamous cell carcinoma or basal cell carcinoma).
   * Patients with a history of severe recurrent or chronic infections, or acute infections requiring systemic treatment with antibiotics, antiviral drugs, antiparasitic drugs, antiamebic drugs, or antifungal drugs within 4 weeks prior to the first dose and during the screening period. Note that superficial skin infections requiring systemic treatment within one week prior to the first dose, if the infection subsides, the patient may be re-screened.
   * Patients with a known or suspected history of immunosuppression, including invasive opportunistic infections such as histoplasmosis, listeriosis, coccidioidomycosis, Pneumocystis pneumonia, and aspergillosis, even if the infection has subsided; or unusually frequent, recurrent, or chronic infections (as judged by the investigator).
   * Patients with significant laboratory abnormalities during the screening period: a) Alanine aminotransferase or aspartate aminotransferase equal to or greater than the upper limit of normal (ULN). b) Total bilirubin equal to or greater than 1.2 times the ULN (note: patients diagnosed with Gilbert's syndrome based on medical history should not be excluded based on this criterion). c) Creatinine and blood urea nitrogen equal to or greater than the ULN.
   * Patients with positive HIV antibodies or syphilis antibodies.
   * Patients who test positive for hepatitis B surface antigen (HBsAg), hepatitis B core antibody, HBV-DNA (detected by polymerase chain reaction), or hepatitis C virus antibody during the screening period. Patients who are positive for hepatitis B core antibody but negative for HBV-DNA may be included, with HBV-DNA monitored every 4 weeks.
   * Pregnant or breastfeeding women, or women who plan to become pregnant or breastfeed during the study; and male patients with a partner planning to become pregnant during the study.
   * Patients with psychiatric disorders, who are unable to provide informed consent and participate in the trial and follow-up.
   * Patients whose toxicity symptoms from prior treatments have not yet resolved are excluded from the trial.
   * Any other conditions deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Time to achieve disease control（DC） | 54 weeks
  The time to achieve disease control and the end of consolidation.
Pemphigus Disease Area Index (PDAl) | 36 week
  Pemphigus Disease Area lndex (PDAl). PDAl activity score cutoffs were defined as 0